CLINICAL TRIAL: NCT03299543
Title: Relationship Among Breath Acetone, Blood Beta-Hydroxybutyrate, and Blood Glucose
Brief Title: Comparison Between Breath Acetone and Blood Beta-Hydroxybutyrate
Status: Completed | Type: Observational
Sponsor: Medamonitor (Industry)
Responsible Party: Sponsor
Other Study IDs: LVL-0717
Record Dates: First submitted 2017-09-22; First posted 2017-10-03 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Ketosis
Keywords: beta-hydroxybutyrate; breath acetone
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Healthy adults: Healthy adults who are able to provide duplicate breath samples and pin-drop blood samples
  Interventions: Device: LEVL (Medamonitor)

INTERVENTIONS:
Device: LEVL (Medamonitor) — Subjects will provide duplicate breath samples to the LEVL device for analysis of breath acetone

SUMMARY:
Subjects will provide blood and breath samples to evaluate the relationship between breath acetone and two blood-bound species: beta-hydroxybutyrate and glucose. Subjects will be asked to provide breath and blood samples at a baseline visit and second optional visit. The two visits will be spaced approximately 3 hours apart.

DETAILED DESCRIPTION:
The LEVL device (Medamonitor, Seattle, WA) provides users a method for assessing their own rate of fat metabolism. The LEVL device measures the concentration acetone in breath that the scientific literature has shown to correlate to the rate of fat metabolism.

Typically, the body uses glucose to meet its metabolic energy requirements. If needed, the body can shift from using glucose to using fat. Many different scenarios can cause this shift. Exercise can deplete accessible carbohydrate stores causing the body to use fats for energy production. Dietary changes that cause fat intake to increase and carbohydrate intake to decrease will alter metabolism to efficiently utilize the change in nutrients. In all of these scenarios, the body reduces it utilization of carbohydrates and, thus, shifts to using fats for energy production.

When the body uses fats as an energy substrate, some of these fat molecules are converted by the liver into acetoacetate, a ketone body. By enzymatic action, acetoacetate (AcAc) can be converted into beta-hydroxybutyrate (BOHB). The same enzyme can generate AcAc from BOHB. Additionally, acetoacetate can convert spontaneously into acetone which, due to its small size and highly water solubility, can readily appear in the breath.

Currently, measurement of BOHB in blood is the gold standard for assessing ketone body concentration, also known as ketosis. BOHB measurement requires an invasive finger puncture to obtain blood and a costly (~$5 / test) assay. Because acetone (BrAce) is a sister ketone body to BOHB, breath acetone may be used to assess ketosis and replace the measurement of BOHB. Data in the scientific literature has shown BrAce to correlate with BOHB. Inferring BOHB concentrations from measurement of BrAce using LEVL is less invasive and is potentially less costly.

Reports have suggested that breath acetone is inversely correlated to blood sugar. However, others have suggested no relationship between the two species. If a relationship does exist, measurement of breath acetone could be used as a surrogate measure for blood sugar, a common assay used by individuals with diabetes.

In this study, subjects will provide blood and breath samples evaluate the relationship between breath acetone and two blood-bound species: BOHB and glucose. Subjects may be asked to provide breath and blood samples at two different times (i.e., visits) spaced approximately 3 hours apart. The second visit is not required for participation in the study (i.e., optional).

ELIGIBILITY:
Inclusion Criteria:

1. Subject must complete the consent process

Exclusion Criteria:

1. Subjects with severe lung disease which would prevent them from providing a breath sample through a large bore tube (e.g., large drinking straw)
2. Subjects with diabetes (Type 1 or Type 2)
3. Subjects who are routinely exposed to paints, paint thinners, gasoline, varnishes, glues, dry cleaning solvents, or industrial cleaning products
4. Daily smoker of cigarettes, e-cigarettes, or marijuana
5. Abstain from alcohol over the prior 24 hours
6. Refrain from consumption of large amounts of garlic

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Breath acetone concentration (ppm) will be compared against blood BOHB concentration (mM). The following methods may be used: summary statistics, plotting, and linear regression. | Through study completion, 4 months
  Both individual and average group measurements will be compared

SECONDARY OUTCOMES:
Breath acetone concentration (ppm) will be compared against blood glucose concentration (mg/dL). The following methods may be used: summary statistics, plotting, and linear regression. | Through study completion, 4 months
  Both individual and average group measurements will be compared
Blood glucose concentration (mg/dL) will be compared against blood BOHB concentration (mM). The following methods may be used: summary statistics, plotting, and linear regression. | Through study completion, 4 months
  Both individual and average group measurements will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Joseph C Anderson, PhD, Principal Investigator — Medamonitor
Locations (1):
- Medamonitor, LLC, Seattle, Washington, United States